CLINICAL TRIAL: NCT00705016
Title: Open-label, Randomized, Controlled Phase I/II Study of Cilengitide to Evaluate the Safety and Efficacy of the Combination of Different Regimens of Cilengitide Added to Cisplatin, 5-FU, and Cetuximab in Subjects With Recurrent/Metastatic Squamous Cell Cancer of the Head and Neck
Brief Title: Cilengitide in Recurrent and/or Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Acronym: ADVANTAGE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 200052-013; 2008-000615-15 (EudraCT Number)
Record Dates: First submitted 2008-06-24; First posted 2008-06-25 (Estimated); Results first posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-03

CONDITIONS: Squamous Cell Cancer
Keywords: Randomized treatment; open-label; controlled; recurrent; metastatic; SCCHN; suitable; for local therapy
MeSH Terms: conditions — Neoplasms, Squamous Cell; Recurrence; Neoplasm Metastasis | interventions — Cilengitide; Cetuximab; Fluorouracil; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cilengitide 2000 mg once weekly+Cetuximab+5-FU+Cisplatin (Experimental)
  Interventions: Drug: Cilengitide 2000 mg once weekly; Drug: Cetuximab; Drug: 5-fluorouracil (5-FU); Drug: Cisplatin
- Cilengitide 2000 mg twice weekly+Cetuximab+5-FU+Cisplatin (Experimental)
  Interventions: Drug: Cilengitide 2000 mg twice weekly; Drug: Cetuximab; Drug: 5-fluorouracil (5-FU); Drug: Cisplatin
- Cetuximab+5-FU+Cisplatin (Active Comparator)
  Interventions: Drug: Cetuximab; Drug: 5-fluorouracil (5-FU); Drug: Cisplatin

INTERVENTIONS:
Drug: Cilengitide 2000 mg once weekly — Cilengitide 500 milligram (mg) will be administered as an intravenous infusion over 60 minutes, daily from Day 1 to 4 of the first week of each 3-week cycle, subsequently followed by 2000 mg dose of cilengitide on Day 8 and 15 of every cycle for a total of 6 cycles (18 weeks) or until PD, unacceptable toxicity or withdrawal for any other reason. After 6 cycles, participants received cilengitide 2000 mg once weekly until PD, unacceptable toxicity or withdrawal for any other reason.
  Arms: Cilengitide 2000 mg once weekly+Cetuximab+5-FU+Cisplatin
Drug: Cilengitide 2000 mg twice weekly — Cilengitide 2000 mg will be administered as an intravenous infusion over 60 minutes, twice weekly on Day 1, 4, 8, 11, 15, and 18 of each 3-week cycle for a total of 6 cycles (18 weeks) or until PD, unacceptable toxicity or withdrawal for any other reason. After 6 cycles, participants will receive cilengitide 2000 mg once weekly until PD, unacceptable toxicity or withdrawal for any other reason.
  Arms: Cilengitide 2000 mg twice weekly+Cetuximab+5-FU+Cisplatin
Drug: Cetuximab — Cetuximab will be administered as 250 milligram per square meter (mg/m^2) as infusion (initial starting dose of 400 mg/m^2) on Day 1, 8 and 15 of each 3-week treatment cycle. Cetuximab will be administered for a total of 6 cycles (18 weeks) or until PD, unacceptable toxicity or withdrawal for any other reason. After 6 cycles, participants received Cetuximab 250 mg/m^2 once weekly until PD, unacceptable toxicity or withdrawal for any other reason.
  Other Names: Erbitux®
Drug: 5-fluorouracil (5-FU) — 5-FU will be administered as an intravenous continuous infusion at a dose of 1000 mg/m^2 daily from Day 1 to 4 of each 3-week treatment cycle. 5-FU will be administered for a total of 6 cycles (18 weeks), or until PD, unacceptable toxicity, or withdrawal for any other reason, whichever occur first.
Drug: Cisplatin — Cisplatin will be administered as an intravenous infusion over 60 minutes, at a dose 100 mg/m^2 on Day 1 of each 3-week treatment cycle. Cisplatin will be administered for a total of 6 cycles (18 weeks), or until PD, unacceptable toxicity, or withdrawal for any other reason, whichever occur first.

SUMMARY:
The purpose of this open-label, randomized, controlled, Phase 1/2 study of the integrin inhibitor cilengitide is to evaluate the safety and efficacy of the combination of different regimens of cilengitide added to cisplatin, 5-fluorouracil (5-FU), and cetuximab in participants with recurrent/metastatic squamous cell carcinoma of the head and neck (SCCHN).

The Phase 1 part was conducted in dedicated study centers. In the Phase 2 part of this trial, cilengitide is administered at two different doses to two experimental groups. The third group will only receive cisplatin, 5-FU and cetuximab. In the Phase 1 part of this trial, the dose of cilengitide in combination with cisplatin, 5-FU and cetuximab was determined.

Cilengitide is an experimental anti-cancer substance interacting with so-called integrins. Integrins are protein molecules that are known to be present on the surface of certain cancer cells. Integrins are also found on certain cells that belong to growing blood vessels (endothelial cells). Integrins potentially facilitate the blood vessels' support of the tumor (angiogenesis) as well as the tumor's growth and further spread throughout the body (metastasis). By inhibiting integrins on the tumor cell surface, cilengitide potentially kills cancer cells, and potentially sensitizes cancer cells to other co-administered therapeutics. By inhibiting integrins on the endothelial cell surface, it potentially inhibits the ingrowth of additional blood vessels towards the tumor.

Cilengitide is given as an intravenous infusion (given by a drip in one vein of your arm). If any unacceptable side effect occurs, treatment with the study drug will be stopped.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of SCCHN
* At least one measurable lesion either by computerized tomography (CT) scan or magnetic resonance imaging (MRI)
* Karnofsky performance status (KPS) of greater than or equal to 70 or eastern cooperative oncology group performance status (ECOG PS) of 0-1 at trial entry

Exclusion Criteria:

* Prior systemic chemotherapy, except if given as part of a multimodal treatment for locally advanced disease, which was completed more than 6 months prior to trial entry
* Surgery (excluding prior diagnostic biopsy) or irradiation within 4 weeks before trial entry
* Nasopharyngeal Carcinoma
* Documented or symptomatic brain or leptomeningeal metastasis
* Previous treatment with epidermal growth factor receptor (EGFR) targeting therapy or signal transduction inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2008-10; Primary Completion 2011-09 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vermorken, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (37):
- Austria (2):
  - Research Site, Salzburg
  - Research Site, Vienna
- Belgium (6):
  - Research Site, Antwerp
  - Research Site, Brussels
  - Research Site, Edegem (Antwerp)
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Namur
- France (7):
  - Research Site, Lille
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Villejuif
- Germany (9):
  - Research Site, Aachen
  - Research Site, Berlin
  - Research Site, Essen
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Jena
  - Research Site, Leipzig
  - Research Site, Rostock
  - Research Site, Stuttgart
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Nyíregyháza
- Italy (3):
  - Research Site, La Spezia
  - Research Site, Milan
  - Research Site, Napoli
- Poland (2):
  - Research Site, Gliwice
  - Research Site, Warsaw
- Spain (3):
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Velencia
- Switzerland (2):
  - Research Site, Basel
  - Research Site, Geneva

REFERENCES:
- [Result] Vermorken JB, Peyrade F, Krauss J, Mesia R, Remenar E, Gauler TC, Keilholz U, Delord JP, Schafhausen P, Erfan J, Brummendorf TH, Iglesias L, Bethe U, Hicking C, Clement PM. Cisplatin, 5-fluorouracil, and cetuximab (PFE) with or without cilengitide in recurrent/metastatic squamous cell carcinoma of the head and neck: results of the randomized phase I/II ADVANTAGE trial (phase II part). Ann Oncol. 2014 Mar;25(3):682-688. doi: 10.1093/annonc/mdu003. PMID 24567516

RESULTS

PARTICIPANT FLOW:
Groups:
- Cilengitide 2000 mg Once Weekly+Cetuximab+5-FU+Cisplatin: Cilengitide 500 milligram (mg) intravenous infusion over 60 minutes, daily from Day 1 to 4 of the first week of each 3-week cycle, subsequently followed by cilengitide 2000 mg once weekly along with cetuximab 250 milligram per square meter (mg/m^2) intravenous infusion (initial starting dose of 400 mg/m^2) once weekly, 5-fluorouracil (5-FU) 1000 mg/m^2 intravenous continuous infusion daily from Day 1 to 4 and cisplatin 100 mg/m^2 intravenous infusion over 60 minutes on Day 1, of each 3-week treatment cycle for a total of 6 cycles (18 weeks) or until progressive disease (PD), unacceptable toxicity or withdrawal for any other reason. After 6 cycles, participants received cilengitide 2000 mg once weekly along with cetuximab 250 mg/m^2 intravenous infusion until PD, unacceptable toxicity or withdrawal for any other reason.
- Cilengitide 2000 mg Twice Weekly+Cetuximab+5-FU+Cisplatin: Cilengitide 2000 mg intravenous infusion over 60 minutes twice weekly along with cetuximab 250 mg/m^2 intravenous infusion (initial starting dose of 400 mg/m^2) once weekly, 5-fluorouracil (5-FU) 1000 mg/m^2 intravenous continuous infusion daily from Day 1 to 4 and cisplatin 100 mg/m^2 intravenous infusion over 60 minutes on Day 1, of each 3-week treatment cycle for a total of 6 cycles (18 weeks) or until PD, unacceptable toxicity or withdrawal for any other reason. After 6 cycles, participants received cilengitide 2000 mg once weekly along with cetuximab 250 mg/m^2 intravenous infusion until PD, unacceptable toxicity or withdrawal for any other reason.
- Cetuximab+5-FU+Cisplatin: Cetuximab 250 mg/m^2 intravenous infusion (initial starting dose of 400 mg/m^2) once weekly along with 5-fluorouracil (5-FU) 1000 mg/m^2 intravenous continuous infusion daily from Day 1 to 4 and cisplatin 100 mg/m^2 intravenous infusion over 60 minutes on Day 1, of each 3-week treatment cycle for a total of 6 cycles (18 weeks) or until PD, unacceptable toxicity or withdrawal for any other reason. After 6 cycles, participants received cetuximab 250 mg/m^2 intravenous infusion until PD, unacceptable toxicity or withdrawal for any other reason.
Period: Overall Study
Arm/Group | Cilengitide 2000 mg Once Weekly+Cetuximab+5-FU+Cisplatin | Cilengitide 2000 mg Twice Weekly+Cetuximab+5-FU+Cisplatin | Cetuximab+5-FU+Cisplatin
Started | 62 | 60 | 62
Completed | 2 | 2 | 4
Not Completed | 60 | 58 | 58
Not completed — Adverse Event | 6 | 11 | 10
Not completed — Death | 5 | 7 | 5
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 4 | 3 | 2
Not completed — Progressive Disease | 33 | 29 | 33
Not completed — Symptomatic Deterioration | 3 | 1 | 1
Not completed — Other | 9 | 6 | 6

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population included all participants who were randomized to trial treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cilengitide 2000 mg Once Weekly+Cetuximab+5-FU+Cisplatin | Cilengitide 2000 mg Twice Weekly+Cetuximab+5-FU+Cisplatin | Cetuximab+5-FU+Cisplatin | Total
Number analyzed (Participants) | 62 | 60 | 62 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] — Out of a total of 62 participants in Cetuximab + 5-FU + Cisplatin group, data for baseline measure (age) was available for 61 participants only.
  years | 59.1 (7.4) | 56.8 (7.9) | 58.6 (8.1) | 58.2 (7.8)
Age, Customized [Number; unit: participants] — Out of a total of 62 participants in Cetuximab + 5-FU + Cisplatin group, data for baseline measure (age) was available for 61 participants only.
  participants
    Less than (<) 65 years | 47 | 48 | 46 | 141
    Greater than or equal to (>=) 65 years | 15 | 12 | 15 | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 6 | 25
  Male | 54 | 49 | 56 | 159
Karnofsky Performance Status [Number; unit: participants] — Karnofsky performance status score ranged from 100 to 0; 100: Normal; 90: Able to Carry on normal Activity; 80: Normal Activity with Effort; Some Signs or Symptoms of Disease; 70: Cares for Self, Unable to Carry on Normal Activity or to Do Active Work; 60: Requires Occasional Assistance but is Able to Care for Most of Needs; 50: Requires Considerable Assistance and Frequent Medical Care; 40: Disabled, Requires Special Care and Assistance; 30: Severely Disabled; Hospitalization Indicated Although Death is Not Imminent; 20: Very Sick; 10: Moribund, Fatal Processes Progressing Rapidly; 0: Death.
  participants
    < 80 (Karnofsky Score) | 7 | 6 | 5 | 18
    >= 80 (Karnofsky Score) | 55 | 54 | 57 | 166
Extent of disease at study entry [Number; unit: participants]
  Recurrence | 30 | 32 | 31 | 93
  Distant Metastasis | 32 | 28 | 31 | 91
Tumor Grade [Number; unit: participants] — Out of a total of 62 participants in Cilengitide 2000 mg once weekly + Cetuximab + 5-FU + Cisplatin group, 60 participants in Cilengitide 2000 mg twice weekly + Cetuximab + 5-FU + Cisplatin group, and 62 participants in Cetuximab + 5-FU + Cisplatin group, data for baseline measure (Tumor grade) was available for 57, 58 and 57 participants only, respectively. Tumor grades were divided in to well or moderately differentiated and poorly differentiated.
  participants
    Well or moderately differentiated | 46 | 39 | 35 | 120
    Poorly differentiated | 11 | 19 | 22 | 52
Site of origin of tumor [Number; unit: participants]
  Oropharynx | 25 | 23 | 21 | 69
  Hypopharynx | 10 | 14 | 14 | 38
  Larynx | 14 | 15 | 13 | 42
  Oral cavity | 11 | 6 | 11 | 28
  Other, including non-classifiable | 2 | 2 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Time: Investigator Read
Description: The PFS is defined as the duration from randomization until radiological progression (based on response evaluation criteria in solid tumors [RECIST] Version 1.0) or death due to any cause. Only deaths within 84 days of last tumor assessment are considered. Participants without event are censored on the date of last tumor assessment. Investigator read is the assessment of all imaging by the treating physician at the local trial site.
Time Frame: Time from randomization to disease progression, death or last tumor assessment, reported between day of first participant randomized, 03 July 2009, until cut-off date (03 September 2011)
Population: Intention-to-treat (ITT) population included all participants who were randomized to trial treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cilengitide 2000 mg Once Weekly+Cetuximab+5-FU+Cisplatin | Cilengitide 2000 mg Twice Weekly+Cetuximab+5-FU+Cisplatin | Cetuximab+5-FU+Cisplatin
Number analyzed (Participants) | 62 | 60 | 62
months | 6.4 [5.4 to 8.7] | 5.6 [4.0 to 6.1] | 5.7 [4.2 to 9.5]
Statistical Analysis 1: Comparison: Cilengitide 2000 mg Once Weekly+Cetuximab+5-FU+Cisplatin vs Cetuximab+5-FU+Cisplatin; Sample size of 177 subjects was estimated such that the treatment group with the best PFS result had a 90% probability of emerging as the one with the smaller observed log Hazard ratio (HR), if there was an underlying difference of 2.2 months between the arms in the median PFS (7.8 months in the best group and 5.6 months in the other 2 groups). It was assumed that the accrual and follow-up time would take 1 year each, and that the drop-out rate was 8%; Test type: Superiority or Other; p = 0.885, Cox proportional hazards model — The Type I error was not taken into account, since the sample size calculation is based on selection theory; Stratification factor: Karnofsky performance status (KPS) <80/>=80; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.67 to 1.59]
Statistical Analysis 2: Comparison: Cilengitide 2000 mg Twice Weekly+Cetuximab+5-FU+Cisplatin vs Cetuximab+5-FU+Cisplatin; Sample size of 177 subjects was estimated such that the treatment group with the best PFS result had a 90% probability of emerging as the one with the smaller observed log HR, if there was an underlying difference of 2.2 months between the arms in the median PFS (7.8 months in the best group and 5.6 months in the other 2 groups). It was assumed that the accrual and follow-up time would take 1 year each, and that the drop-out rate was 8%; Test type: Superiority or Other; p = 0.054, Cox proportional hazards model — The Type I error was not taken into account, since the sample size calculation is based on selection theory; Stratification factor: Karnofsky performance status (KPS) <80/>=80; Hazard Ratio (HR) = 1.55, 95% CI 2-sided [0.99 to 2.43]

2. Secondary Outcome: Overall Survival (OS) Time
Description: The OS time is defined as the time from randomization to death. Participants without event are censored at the last date known to be alive or at the clinical cut-off date, whichever is earlier.
Time Frame: Time from randomization to death, reported between day of first participant randomized, 03 July 2009, until cut-off date (03 September 2011)
Population: ITT population included all participants who were randomized to trial treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cilengitide 2000 mg Once Weekly+Cetuximab+5-FU+Cisplatin | Cilengitide 2000 mg Twice Weekly+Cetuximab+5-FU+Cisplatin | Cetuximab+5-FU+Cisplatin
Number analyzed (Participants) | 62 | 60 | 62
months | 12.4 [9.4 to 14.5] | 10.6 [9.0 to 14.8] | 11.6 [7.1 to 16.4]
Statistical Analysis 1: Comparison: Cilengitide 2000 mg Once Weekly+Cetuximab+5-FU+Cisplatin vs Cetuximab+5-FU+Cisplatin; Test type: Superiority or Other; p = 0.800, Cox proportional hazards model — Secondary analyses of efficacy were performed to support the results of the primary analysis and considered as purely exploratory and no adjustment for multiplicity has been done; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.61 to 1.47]
Statistical Analysis 2: Comparison: Cilengitide 2000 mg Twice Weekly+Cetuximab+5-FU+Cisplatin vs Cetuximab+5-FU+Cisplatin; Test type: Superiority or Other; p = 0.878, Cox proportional hazards model; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.66 to 1.63]

3. Secondary Outcome: Best Overall Response (BOR) Rate
Description: The BOR rate is defined as the percentage of the participants having achieved confirmed complete response (CR) or partial response (PR) as the best overall response according to radiological assessments (based on RECIST Version 1.0).
Time Frame: Evaluations will be performed every 6 weeks until progression reported between day of first participant randomized, 03 July 2009, until cut-off date (03 September 2011)
Population: ITT population included all participants who were randomized to trial treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cilengitide 2000 mg Once Weekly+Cetuximab+5-FU+Cisplatin | Cilengitide 2000 mg Twice Weekly+Cetuximab+5-FU+Cisplatin | Cetuximab+5-FU+Cisplatin
Number analyzed (Participants) | 62 | 60 | 62
percentage of participants | 46.8 [34.0 to 59.9] | 26.7 [16.1 to 39.7] | 35.5 [23.7 to 48.7]
Statistical Analysis 1: Comparison: Cilengitide 2000 mg Once Weekly+Cetuximab+5-FU+Cisplatin vs Cetuximab+5-FU+Cisplatin; Test type: Superiority or Other; p = 0.205, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.595, 95% CI 2-sided [0.776 to 3.276]
Statistical Analysis 2: Comparison: Cilengitide 2000 mg Twice Weekly+Cetuximab+5-FU+Cisplatin vs Cetuximab+5-FU+Cisplatin; Test type: Superiority or Other; p = 0.317, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.671, 95% CI 2-sided [0.307 to 1.465]

4. Secondary Outcome: Disease Control Rate
Description: The disease control rate is defined as the percentage of participants having achieved confirmed CR, PR or stable disease (SD) as best overall response according to radiological assessments (based on RECIST Version 1.0).
Time Frame: as for outcome 3
Population: ITT population included all participants who were randomized to trial treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cilengitide 2000 mg Once Weekly+Cetuximab+5-FU+Cisplatin | Cilengitide 2000 mg Twice Weekly+Cetuximab+5-FU+Cisplatin | Cetuximab+5-FU+Cisplatin
Number analyzed (Participants) | 62 | 60 | 62
percentage of participants | 85.5 [74.2 to 93.1] | 73.3 [60.3 to 83.9] | 80.6 [68.6 to 89.6]
Statistical Analysis 1: Comparison: Cilengitide 2000 mg Once Weekly+Cetuximab+5-FU+Cisplatin vs Cetuximab+5-FU+Cisplatin; Test type: Superiority or Other; p = 0.476, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.396, 95% CI 2-sided [0.551 to 3.539]
Statistical Analysis 2: Comparison: Cilengitide 2000 mg Twice Weekly+Cetuximab+5-FU+Cisplatin vs Cetuximab+5-FU+Cisplatin; Test type: Superiority or Other; p = 0.347, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.668, 95% CI 2-sided [0.287 to 1.555]

5. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF is defined as the time from randomization to date of the first occurrence of; progression, discontinuation of treatment due to progression or adverse event, start of new anticancer therapy, withdrawal of consent, or death (within 84 days of last tumor assessment). Participants without event are censored on the date of last tumor assessment.
Time Frame: as for outcome 1
Population: ITT population included all participants who were randomized to trial treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cilengitide 2000 mg Once Weekly+Cetuximab+5-FU+Cisplatin | Cilengitide 2000 mg Twice Weekly+Cetuximab+5-FU+Cisplatin | Cetuximab+5-FU+Cisplatin
Number analyzed (Participants) | 62 | 60 | 62
months | 5.6 [4.2 to 6.9] | 4.5 [2.9 to 5.6] | 4.3 [3.8 to 7.3]
Statistical Analysis 1: Comparison: Cilengitide 2000 mg Once Weekly+Cetuximab+5-FU+Cisplatin vs Cetuximab+5-FU+Cisplatin; Test type: Superiority or Other; p = 0.294, Cox proportional hazards model — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.84 to 1.81]
Statistical Analysis 2: Comparison: Cilengitide 2000 mg Twice Weekly+Cetuximab+5-FU+Cisplatin vs Cetuximab+5-FU+Cisplatin; Test type: Superiority or Other; p = 0.007, Cox proportional hazards model — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.73, 95% CI 2-sided [1.16 to 2.57]

6. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from the first assessment of CR or PR until the date of the first occurrence of progressive disease (PD), or until the date of death.
Time Frame: Time from first assessment of CR or PR until PD, death or last tumor assessment, reported between day of first participant randomized, 03 July 2009, until cut-off date (03 September 2011)
Population: ITT population included all participants who were randomized to trial treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cilengitide 2000 mg Once Weekly+Cetuximab+5-FU+Cisplatin | Cilengitide 2000 mg Twice Weekly+Cetuximab+5-FU+Cisplatin | Cetuximab+5-FU+Cisplatin
Number analyzed (Participants) | 62 | 60 | 62
months | 5.8 [4.5 to 7.5] | 4.1 [3.1 to 4.4] | 6.4 [4.2 to 9.7]
Statistical Analysis 1: Comparison: Cilengitide 2000 mg Once Weekly+Cetuximab+5-FU+Cisplatin vs Cetuximab+5-FU+Cisplatin; Test type: Superiority or Other; p = 0.391, Cox proportional hazards model — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [0.71 to 2.39]
Statistical Analysis 2: Comparison: Cilengitide 2000 mg Twice Weekly+Cetuximab+5-FU+Cisplatin vs Cetuximab+5-FU+Cisplatin; Test type: Superiority or Other; p = 0.007, Cox proportional hazards model — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 2.60, 95% CI 2-sided [1.30 to 5.21]

7. Secondary Outcome: Safety - Number of Participants Experiencing Any Adverse Event
Description: Please refer to Adverse Events section for details of individual serious adverse events and other adverse events
Time Frame: as for outcome 6
Population: Safety population included all participants who were administered any dose of the trial medication, that is, cilengitide, cisplatin, 5-FU, or cetuximab.
Measure: Number; unit: participants
Arm/Group | Cilengitide 2000 mg Once Weekly+Cetuximab+5-FU+Cisplatin | Cilengitide 2000 mg Twice Weekly+Cetuximab+5-FU+Cisplatin | Cetuximab+5-FU+Cisplatin
Number analyzed (Participants) | 61 | 59 | 62
participants | 61 | 59 | 61

ADVERSE EVENTS:
Time Frame: Time from first dose up to 28 days after last dose of study treatment, reported between day of first patient randomized, 01 October 2008, until cut off date, 03 September 2011
Arm/Group | Cilengitide 2000 mg Once Weekly+Cetuximab+5-FU+Cisplatin | Cilengitide 2000 mg Twice Weekly+Cetuximab+5-FU+Cisplatin | Cetuximab+5-FU+Cisplatin
Serious Adverse Events (participants affected / at risk) | 41/61 | 45/59 | 44/62
Other Adverse Events (participants affected / at risk) | 61/61 | 57/59 | 61/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cilengitide 2000 mg Once Weekly+Cetuximab+5-FU+Cisplatin (N=61) | Cilengitide 2000 mg Twice Weekly+Cetuximab+5-FU+Cisplatin (N=59) | Cetuximab+5-FU+Cisplatin (N=62)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 4 (6) | 5 (5)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Duodenal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large Intestine Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenic Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophageal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tongue Necrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 5 (5) | 5 (6)
Sepsis (Infections and infestations) | 3 (4) | 0 (0) | 2 (2)
Device Related Infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Escherichia Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Pulmonary Sepsis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Catheter Site Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dermatitis Infected (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis Infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral Fungal Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
General Physical Health Deterioration (General disorders) | 3 (3) | 4 (4) | 2 (3)
Pyrexia (General disorders) | 2 (2) | 4 (4) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1) | 3 (3)
Device Dislocation (General disorders) | 0 (0) | 2 (3) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 0 (0) | 0 (0)
Face Oedema (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Thrombosis In Device (General disorders) | 1 (1) | 1 (1) | 0 (0)
Catheter Site Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Device Leakage (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperpyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Performance Status Decreased (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 6 (7) | 5 (7)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (5) | 6 (6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (6) | 1 (2) | 9 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 6 (11) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 4 (5) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary Artery Thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 2 (2) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Axillary Vein Thrombosis (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Arterial Rupture (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis Obliterans (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Jugular Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 3 (3) | 3 (3) | 1 (1)
Cerebral Infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depressed Level Of Consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Blood Creatinine Increased (Investigations) | 0 (0) | 1 (2) | 2 (2)
Blood Amylase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood Creatine Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Glomerular Filtration Rate Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 2 (2) | 2 (2) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Gastrostomy Failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ototoxicity (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Paraneoplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
Infected Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Retinal Artery Occlusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal Artery Thrombosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual Acuity Reduced (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cilengitide 2000 mg Once Weekly+Cetuximab+5-FU+Cisplatin (N=61) | Cilengitide 2000 mg Twice Weekly+Cetuximab+5-FU+Cisplatin (N=59) | Cetuximab+5-FU+Cisplatin (N=62)
Nausea (Gastrointestinal disorders) | 36 (98) | 31 (78) | 40 (137)
Stomatitis (Gastrointestinal disorders) | 27 (85) | 28 (77) | 30 (83)
Vomiting (Gastrointestinal disorders) | 28 (66) | 24 (55) | 28 (96)
Diarrhoea (Gastrointestinal disorders) | 23 (45) | 27 (60) | 24 (65)
Constipation (Gastrointestinal disorders) | 23 (43) | 22 (37) | 24 (36)
Dysphagia (Gastrointestinal disorders) | 5 (11) | 7 (10) | 8 (12)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 3 (4) | 11 (16)
Abdominal Pain Upper (Gastrointestinal disorders) | 6 (9) | 5 (5) | 4 (6)
Abdominal Pain (Gastrointestinal disorders) | 7 (9) | 7 (9) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 3 (3) | 2 (2) | 4 (4)
Odynophagia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 4 (4)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 4 (5)
Gastritis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 22 (54) | 22 (99) | 27 (91)
Dry Skin (Skin and subcutaneous tissue disorders) | 15 (35) | 13 (19) | 11 (18)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 11 (29) | 11 (30) | 11 (34)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (19) | 9 (13) | 11 (12)
Skin Fissures (Skin and subcutaneous tissue disorders) | 10 (32) | 9 (19) | 12 (22)
Erythema (Skin and subcutaneous tissue disorders) | 9 (22) | 2 (2) | 5 (5)
Acne (Skin and subcutaneous tissue disorders) | 6 (8) | 4 (8) | 5 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (11) | 3 (8) | 3 (6)
Nail Disorder (Skin and subcutaneous tissue disorders) | 3 (6) | 7 (13) | 1 (4)
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 5 (11) | 3 (6) | 2 (3)
Exfoliative Rash (Skin and subcutaneous tissue disorders) | 4 (27) | 3 (6) | 1 (1)
Fatigue (General disorders) | 20 (47) | 24 (62) | 24 (65)
Asthenia (General disorders) | 21 (80) | 7 (28) | 17 (61)
Pyrexia (General disorders) | 14 (23) | 13 (17) | 18 (39)
Oedema Peripheral (General disorders) | 5 (13) | 11 (26) | 10 (17)
Face Oedema (General disorders) | 1 (1) | 3 (3) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 28 (63) | 24 (108) | 29 (80)
Anaemia (Blood and lymphatic system disorders) | 22 (57) | 16 (45) | 22 (65)
Leukopenia (Blood and lymphatic system disorders) | 16 (38) | 15 (52) | 12 (39)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (24) | 15 (33) | 14 (30)
Lymphopenia (Blood and lymphatic system disorders) | 5 (8) | 2 (6) | 3 (13)
Normochromic Normocytic Anaemia (Blood and lymphatic system disorders) | 1 (6) | 3 (4) | 5 (5)
Decreased Appetite (Metabolism and nutrition disorders) | 20 (37) | 15 (42) | 18 (45)
Hypokalaemia (Metabolism and nutrition disorders) | 19 (41) | 15 (50) | 15 (37)
Hypomagnesaemia (Metabolism and nutrition disorders) | 17 (36) | 13 (55) | 14 (38)
Hypocalcaemia (Metabolism and nutrition disorders) | 6 (13) | 8 (25) | 9 (32)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (19) | 7 (21) | 4 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 6 (6) | 3 (4) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 3 (3) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 5 (7)
Paronychia (Infections and infestations) | 7 (10) | 4 (10) | 6 (11)
Folliculitis (Infections and infestations) | 6 (10) | 6 (16) | 4 (8)
Pneumonia (Infections and infestations) | 4 (4) | 5 (5) | 2 (2)
Device Related Infection (Infections and infestations) | 5 (6) | 3 (4) | 1 (1)
Oral Candidiasis (Infections and infestations) | 4 (8) | 3 (4) | 1 (1)
Infection (Infections and infestations) | 2 (4) | 3 (3) | 3 (3)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (4) | 2 (4)
Oral Fungal Infection (Infections and infestations) | 0 (0) | 3 (4) | 3 (7)
Weight Decreased (Investigations) | 12 (22) | 10 (12) | 12 (15)
Haemoglobin Decreased (Investigations) | 8 (39) | 9 (35) | 7 (22)
Blood Creatinine Increased (Investigations) | 6 (6) | 8 (18) | 7 (13)
Platelet Count Decreased (Investigations) | 4 (14) | 5 (8) | 6 (19)
Neutrophil Count Decreased (Investigations) | 7 (26) | 3 (7) | 4 (11)
White Blood Cell Count Decreased (Investigations) | 7 (32) | 2 (18) | 4 (19)
Dizziness (Nervous system disorders) | 8 (18) | 9 (20) | 6 (14)
Headache (Nervous system disorders) | 8 (13) | 4 (4) | 5 (6)
Paraesthesia (Nervous system disorders) | 6 (17) | 4 (7) | 5 (7)
Peripheral Sensory Neuropathy (Nervous system disorders) | 4 (10) | 7 (15) | 3 (12)
Dysgeusia (Nervous system disorders) | 4 (5) | 2 (2) | 5 (6)
Neuropathy Peripheral (Nervous system disorders) | 6 (14) | 1 (1) | 2 (4)
Polyneuropathy (Nervous system disorders) | 5 (5) | 2 (2) | 2 (4)
Syncope (Nervous system disorders) | 2 (2) | 3 (4) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (17) | 9 (11) | 10 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (14) | 12 (17) | 6 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 9 (13) | 4 (10)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 5 (8) | 6 (8)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (2) | 4 (8)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 7 (7) | 3 (4)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (8) | 4 (5)
Neck Pain (Musculoskeletal and connective tissue disorders) | 4 (7) | 3 (4) | 2 (2)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 0 (0)
Hypertension (Vascular disorders) | 7 (11) | 6 (11) | 8 (14)
Hypotension (Vascular disorders) | 6 (8) | 8 (11) | 4 (7)
Phlebitis (Vascular disorders) | 2 (2) | 3 (4) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 3 (7) | 5 (9) | 4 (4)
Deafness (Ear and labyrinth disorders) | 5 (6) | 3 (4) | 4 (4)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 5 (6) | 3 (9)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 4 (4) | 1 (1)
Conjunctivitis (Eye disorders) | 8 (9) | 3 (5) | 10 (13)
Insomnia (Psychiatric disorders) | 4 (6) | 7 (8) | 6 (6)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1) | 4 (4)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 4 (7)
Dysuria (Renal and urinary disorders) | 2 (2) | 3 (4) | 1 (3)
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 6 (13) | 6 (11)
Drug Hypersensitivity (Immune system disorders) | 3 (3) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less